CLINICAL TRIAL: NCT03399786
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Evinacumab in Patients With Homozygous Familial Hypercholesterolemia
Brief Title: Efficacy and Safety of Evinacumab in Patients With Homozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R1500-CL-1629; 2017-001388-19 (EudraCT Number)
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: HoFH
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — evinacumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- evinacumab (Experimental)
  Interventions: Drug: evinacumab
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: evinacumab — IV administration of evinacumab
  Other Names: REGN1500
  Arms: evinacumab
Drug: Placebo — IV administration of placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by evinacumab intravenously (IV) in comparison to placebo after 24 weeks in patients with homozygous familial hypercholesterolemia (HoFH). The secondary objectives of the study are to evaluate the effect of evinacumab IV on other lipid parameters, evaluate the effect of evinacumab on LDL-C goal attainment, assess the effect of evinacumab on eligibility for apheresis (using German and US apheresis criteria), evaluate the safety and tolerability of evinacumab in patients with HoFH, assess the pharmacokinetics (PK) of evinacumab in patients with HoFH and evaluate the potential development of anti-evinacumab antibodies.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of functional HoFH
2. If undergoing LDL apheresis, must have initiated LDL apheresis at least 3 months prior to screening and must have been on a stable weekly or every other week schedule and/or stable settings for at least 8 weeks
3. Willing to consistently maintain his/her usual low fat or heart-healthy diet for the duration of the study

Key Exclusion Criteria:

1. LDL-C level <70 mg/dL (1.81 mmol/L) at the screening visit
2. Background medical Lipid Modifying Therapy (LMT) (if applicable) that has not been stable before the screening visit
3. Lipid-apheresis schedule /apheresis settings (if applicable) that have not been stable for at least 8 weeks before the screening visit
4. Use of nutraceuticals or over-the-counter therapies known to affect lipids, at a dose/amount that has not been stable for at least 4 weeks prior to the screening visit
5. Presence of any clinically significant uncontrolled endocrine disease known to influence serum lipids or lipoproteins
6. Newly diagnosed (within 3 months prior to randomization visit) diabetes mellitus or poorly controlled (HbA1c >9%) diabetes
7. History of a MI, unstable angina leading to hospitalization, coronary artery bypass graft surgery, percutaneous coronary intervention, uncontrolled cardiac arrhythmia, carotid surgery or stenting, stroke, transient ischemic attack, valve replacement surgery, carotid revascularization, endovascular procedure or surgical intervention for peripheral vascular disease within 3 months prior to the screening visit
8. Pregnant or breastfeeding women
9. Sexually active women of child bearing potential (WOCBP), who are unwilling to practice a highly effective birth control method prior to the initial dose, during the study, and for 24 weeks after the last dose of study drug
10. Men who are sexually active with women of child bearing potential (WOCBP) and are unwilling to consistently use condoms during the study drug treatment period and for 24 weeks after the last dose of study drug regardless of vasectomy status

Note: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (30):
- United States (6):
  - Regeneron Research Site, Boca Raton, Florida
  - Regeneron Research Site, Boston, Massachusetts
  - Regeneron Research Site, New York, New York
  - Regeneron Research Site, Cincinnati, Ohio
  - Regeneron Research Site, Portland, Oregon
  - Regeneron Research Site, Dallas, Texas
- Australia (2):
  - Regeneron Research Site, Camperdown, New South Wales
  - Regeneron Research Site, Perth, Western Australia
- Regeneron Research Site, Innsbruck, Austria
- Canada (2):
  - Regeneron Research Site, Chicoutimi, Quebec
  - Regeneron Research Site, Québec, Quebec
- France (2):
  - Regeneron Research Site, Paris, Cedex
  - Regeneron Research Site, Marseille
- Greece (2):
  - Regeneron Research Site, Ioannina, Ioannina
  - Regeneron Research Site, Athens
- Regeneron Research Site # 2, Napoli, Italy
- Japan (6):
  - Regeneron Research Site, Kurume, Fukuoka
  - Regeneron Research Site, Nishinomiya, Hyōgo
  - Regeneron Research Site, Kanazawa, Ishikawa-ken
  - Regeneron Research Site #3, Suita, Osaka
  - Regeneron Research Site, Suita, Osaka
  - Regeneron Research Site, Osaka
- Netherlands (2):
  - Regeneron Research Site, Amsterdam
  - Regeneron Research Site, Rotterdam
- Regeneron Research Site, Parktown, Johannesburg, South Africa
- Ukraine (5):
  - Regeneron Research Site, Ivano-Frankivsk
  - Regeneron Research Site, Kharkiv
  - Regeneron Research Site #2, Kharkiv
  - Regeneron Research Site #2, Kyiv
  - Regeneron Research Site, Kyiv

REFERENCES:
- [Derived] Iannuzzo G, Calcaterra I, Gentile M, Stanzione C, De Ruberto F, Di Taranto MD, Fortunato G, Di Minno M. Evinacumab for Homozygous Familial Hypercholesterolemia: The Italian Cohort of the ELIPSE HoFH Study. Adv Ther. 2025 May;42(5):2465-2479. doi: 10.1007/s12325-025-03160-4. Epub 2025 Apr 2. PMID 40169529
- [Derived] Raal FJ, Rosenson RS, Reeskamp LF, Hovingh GK, Kastelein JJP, Rubba P, Ali S, Banerjee P, Chan KC, Gipe DA, Khilla N, Pordy R, Weinreich DM, Yancopoulos GD, Zhang Y, Gaudet D; ELIPSE HoFH Investigators. Evinacumab for Homozygous Familial Hypercholesterolemia. N Engl J Med. 2020 Aug 20;383(8):711-720. doi: 10.1056/NEJMoa2004215. PMID 32813947

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 30 centers that enrolled participants in 11 countries in Europe, Asia, North America, and Australia. Randomization was stratified by apheresis treatment status and by region (Japan, Rest of the World [ROW]).
Pre-assignment Details: A total of 75 participants were screened and 65 participants randomized. There were 10 participants that were considered screen failures.
Groups:
- Placebo IV Q4W (DBTP): Participants received IV infusion of placebo matched to evinacumab every 4 weeks (Q4W) from day 1 to week 20 in the double-blind treatment period (DBTP).
- Evinacumab 15 mg/kg (DBTP): Participants received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from day 1 to week 20 in the double-blind treatment period (DBTP).
- Placebo IV Q4W (OLTP): All participants in the placebo arm who completed the double-blind treatment period (DBTP) received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from week 24 to week 44 in the open-label treatment period (OLTP).
- Evinacumab 15 mg/kg (OLTP): All participants in the evinacumab arm who completed the double-blind treatment period (DBTP) received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from week 24 to week 44 in the open-label treatment period (OLTP).
Period: Double-blind Treatment Period (DBTP)
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP) | Placebo IV Q4W (OLTP) | Evinacumab 15 mg/kg (OLTP)
Started | 22 | 43 | 0 | 0
Completed | 21 | 43 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Open-label Treatment Period (OLTP)
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP) | Placebo IV Q4W (OLTP) | Evinacumab 15 mg/kg (OLTP)
Started | 0 | 0 | 20 (One participant from the placebo group received evinacumab during the DBTP) | 44
Completed | 0 | 0 | 19 | 43
Not Completed | 0 | 0 | 1 | 1
Not completed — Noncompliance with protocol by the participant | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo IV Q4W: Participants received IV infusion of placebo matched to evinacumab every 4 weeks (Q4W) from day 1 to week 20 in the double-blind treatment period (DBTP). All participants who completed the double-blind treatment period received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from week 24 to week 44 in the open-label treatment period (OLTP).
- Evinacumab 15 mg/kg IV Q4W: Participants received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from day 1 to week 20 in the double-blind treatment period (DBTP). All participants who completed the double-blind treatment period received IV infusion of evinacumab at a dose of 15 mg/kg Q4W from week 24 to week 44 in the open-label treatment period (OLTP).
- Total: Total of all reporting groups
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W | Total
Number analyzed (Participants) | 22 | 43 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.7 (11.52) | 44.3 (16.78) | 41.7 (15.54)
Age, Customized [Number; unit: Participants]
  ≥12 years to <18 years of age | 1 | 1 | 2
  ≥18 years to <45 years of age | 16 | 23 | 39
  ≥45 years to <65 years of age | 5 | 11 | 16
  ≥65 years to <75 years of age | 0 | 7 | 7
  ≥75 years of age | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 24 | 35
  Male | 11 | 19 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 38 | 58
  Unknown or Not Reported | 1 | 4 | 5
Race [Count of Participants; unit: Participants]
  White | 17 | 31 | 48
  Black or African American | 0 | 2 | 2
  Asian | 4 | 6 | 10
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Not Reported | 0 | 2 | 2
  Other | 1 | 2 | 3
Calculated Low-density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: Milligrams per Deciliter (mg/dL)] | 246.5 (153.71) | 259.5 (172.40) | 255.1 (165.21)
Apolipoprotein B (Apo B) [Mean (Standard Deviation); unit: mg/dL] | 175.9 (98.76) | 169.1 (82.75) | 171.4 (87.78)
Non-high-density Lipoprotein Cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 269.9 (157.81) | 281.9 (172.61) | 277.8 (166.60)
Total Cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 315.9 (150.44) | 325.6 (170.76) | 322.3 (163.05)
Lipoprotein A (Lp[a]) [Mean (Standard Deviation); unit: Nanomoles per Liter (nmol/L)] | 103.4 (109.43) | 111.3 (114.40) | 108.7 (111.95)
Fasting Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 144.1 (144.54) | 113.1 (68.39) | 123.6 (100.71)
Apolipoprotein CIII (Apo CIII) [Mean (Standard Deviation); unit: mg/dL] | 9.7 (5.23) | 9.2 (4.00) | 9.39 (4.42)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 24 (Intent-to-Treat [ITT] Estimand)
Description: Percent change was calculated as 100x(calculated LDL-C value at Week 24 - calculated LDL-C value at baseline)/calculated LDL-C value at baseline. The baseline LDL-C value was the last calculated LDL-C value obtained before the first dose of double-blind-study drug. The calculated LDL-C at week 24 was the LDL-C value obtained within the week 24 efficacy analysis window, regardless of adherence to treatment and subsequent therapies (intent-to-treat [ITT] estimand). The ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percent Change | 1.9 (6.5) [lower limit 6.5] | -47.1 (4.6) [lower limit 4.6]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; Confidence interval (CI) with p-value was based on-treatment group difference of least squares (LS) means using mixed-effect model repeat measurement (MMRM), randomization strata, treatment/strata/baseline value-by-time point interaction and continuous fixed covariates of baseline calculated LDL-C value; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeat Measure (MMRM); Least Squares (LS) Mean Difference = -49.0, 95% CI 2-sided [-65.0 to -33.1], Standard Error of Mean 8.0

2. Secondary Outcome: Percent Change in Apolipoprotein B (Apo B) From Baseline to Week 24 (ITT Estimand)
Description: Percent change in Apo B from baseline at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percent Change | -4.5 (4.8) [lower limit 4.8] | -41.4 (3.3) [lower limit 3.3]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; A 2-sided hierarchical testing procedure was used for the secondary endpoints in a pre-specified order to control type I error. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level. CI with p-value was based on-treatment group difference of LS means using MMRM, randomization strata, treatment/strata/baseline value-by-time point interaction and continuous fixed covariates of baseline calculated Apo B value; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeat Measure (MMRM); Least Squares (LS) Mean Difference = -36.9, 95% CI 2-sided [-48.6 to -25.2], Standard Error of Mean 5.9

3. Secondary Outcome: Percent Change in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Week 24 (ITT Estimand)
Description: Percent change from baseline in non-HDL-C at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percent Change | 2.0 (5.4) [lower limit 5.4] | -49.7 (3.8) [lower limit 3.8]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; A 2-sided hierarchical testing procedure was used for the secondary endpoints in a pre-specified order to control type I error. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level. CI with p-value was based on-treatment group difference of LS means using MMRM, randomization strata, treatment/strata/baseline value-by-time point interaction and continuous fixed covariates of baseline calculated non-HDL-C value; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeat Measure (MMRM); Least Squares (LS) Mean Difference = -51.7, 95% CI 2-sided [-64.8 to -38.5], Standard Error of Mean 6.6

4. Secondary Outcome: Percent Change in Total Cholesterol (TC) From Baseline to Week 24 (ITT Estimand)
Description: Percent change in TC from baseline at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percent Change | 1.0 (4.2) [lower limit 4.2] | -47.4 (3.0) [lower limit 3.0]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; A 2-sided hierarchical testing procedure was used for the secondary endpoints in a pre-specified order to control type I error. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level. CI with p-value was based on-treatment group difference of LS means using MMRM, randomization strata, treatment/strata/baseline value-by-time point interaction and continuous fixed covariates of baseline calculated TC value; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeat Measure (MMRM); Least Squares (LS) Mean Difference = -48.4, 95% CI 2-sided [-58.7 to -38.1], Standard Error of Mean 5.1

5. Secondary Outcome: Percentage of Participants With ≥30% Reduction in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24 (ITT Estimand)
Description: Percentage of participants who achieved reduction in calculated LDL-C ≥30% at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: At Week 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percentage of Participants | 18.2 | 83.7
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; A 2-sided hierarchical testing procedure was used for secondary endpoints in pre-specified order to control type I error.Testing sequence continued only when previous endpoint was statistically significant at 0.05.Multiple imputation addressed missing data at week 24.Combined estimate for odds ratio obtained by Rubin's formulae.Logistic regression models stratified by randomized strata include fixed categorical effect of treatment group & continuous fixed covariate of baseline calculated LDL-C; Test type: Superiority — A 2-step multiple imputation method addressed missing values (seeds = 1629 & 9261 with number of imputations = 100 in first and number of imputation=1 in second step); p < 0.0001, Logistic Regression Models Analyses; Odds Ratio (OR) = 25.2, 95% CI 2-sided [5.7 to 110.5]

6. Secondary Outcome: Percentage of Participants With ≥50% Reduction in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24 (ITT Estimand)
Description: Percentage of participants who achieved reduction in calculated LDL-C ≥ 50% at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: At Week 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percentage of Participants | 4.5 | 55.8
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0028, Logistic Regression Models Analyses; Odds Ratio (OR) = 24.2, 95% CI 2-sided [3.0 to 195.6]

7. Secondary Outcome: Absolute Change in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 24 (ITT Estimand)
Description: Absolute change in calculated LDL-C from baseline at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: Milligrams per Deciliter (mg/dL)
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Milligrams per Deciliter (mg/dL) | -2.6 (17.6) [lower limit 17.6] | -134.7 (12.4) [lower limit 12.4]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; A 2-sided hierarchical testing procedure was used for the secondary endpoints in a pre-specified order to control type I error. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level. CI with p-value was based on-treatment group difference of LS means using MMRM, randomization strata, treatment/strata/baseline value-by-time point interaction and continuous fixed covariates of baseline calculated LDL-C value; Test type: Superiority; p < 0.0001, Mixed-effect Model Repeat Measure (MMRM); Least Squares (LS) Mean Difference = -132.1, 95% CI 2-sided [-175.3 to -88.9], Standard Error of Mean 21.5

8. Secondary Outcome: Percentage of Participants Who Met United States (US) Apheresis Eligibility Criteria at Week 24 (ITT Estimand)
Description: US apheresis eligibility criteria included participants who had inadequate response to diet and LMTs after 6 months of treatment and with functional Homozygous familial hypercholesterolemia (HoFH) or Heterozygous familial hypercholesterolemia (HeFH) (with 0-1 risk factor) with LDL-C ≥ 300 mg/dL (7.77 mmol/L). Percentage of participants who met US apheresis eligibility criteria at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: At Week 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percentage of Participants | 22.7 | 7.0
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; A 2-sided hierarchical testing procedure was used for the secondary endpoints in a pre-specified order to control type I error. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level. Combined estimate for odds ratio was obtained by using Rubin's formulae. Logistic regression models stratified the fixed categorical effect of treatment group and the continuous fixed covariate of baseline calculated LDL-C value; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0845, Logistic Regression Models Analyses; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0 to 1.3]

9. Secondary Outcome: Percentage of Participants With Low-Density Lipoprotein Cholesterol (LDL-C) <100 Milligrams Per Deciliter (mg/dL) (2.59 Millimoles Per Liter [mmol/L]) at Week 24 (ITT Estimand)
Description: Percentage of participants with LDL-C value <100 mg/dL (2.59 mmol/L) in the DBTP at Week 24 was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analysed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: At Week 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percentage of Participants | 22.7 | 46.5
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; [analysis description as in outcome 8, analysis 1]; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0203, Logistic Regression Models Analyses — The p-value is nominal for descriptive purpose only due to statistical hypothesis testing terminated previously; Odds Ratio (OR) = 5.7, 95% CI 2-sided [1.3 to 24.9]

10. Secondary Outcome: Percentage of Participants Who Met European Union (EU) Apheresis Eligibility Criteria at Week 24 (ITT Estimand)
Description: EU apheresis eligibility criteria included participants who had inadequate response to diet and Lipid modifying therapies (LMTs) after 3 months of treatment, Primary prevention: Participants with Familial hypercholesterolemia (FH) with LDL-C >160 mg/dL (4.2 mmol/L) and Cardiovascular (CV) events in close relatives. Secondary prevention: Participants with progressive CV events with LDL-C > 120 to 130 mg/dL (3.1-3.4 mmol/L). Percentage of participants who met EU apheresis eligibility criteria at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: At Week 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percentage of Participants | 77.3 | 32.6
Statistical Analysis 1: Comparison: Placebo IV Q4W vs Evinacumab 15 mg/kg IV Q4W; [analysis description as in outcome 8, analysis 1]; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0004, Logistic Regression Models Analysis — The p-value is nominal for descriptive purpose only due to statistical hypothesis testing terminated previously; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0.0 to 0.3]

11. Secondary Outcome: Percentage of Participants With Calculated Low-Density Lipoprotein Cholesterol (LDL-C) <70 mg/dL (1.81 mmol/L) at Week 24 (ITT Estimand)
Description: Percentage of participants with LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: At Week 24
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percentage of Participants | 4.5 | 27.9

12. Secondary Outcome: Percent Change in Fasting Triglycerides (TG) From Baseline to Week 24 (ITT Estimand)
Description: Percent change from baseline in TG at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percent Change | -4.6 (7.0) [lower limit 7.0] | -55.0 (3.1) [lower limit 3.1]

13. Secondary Outcome: Percent Change in Lipoprotein A (Lp[a]) From Baseline to Week 24 (ITT Estimand)
Description: Percent change in Lp(a) from baseline at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percent Change | -3.6 (5.8) [lower limit 5.8] | -5.5 (4.0) [lower limit 4.0]

14. Secondary Outcome: Absolute Change in Apolipoprotein B (Apo B) From Baseline to Week 24 (ITT Estimand)
Description: Absolute change in Apo B from baseline at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
mg/dL | -8.0 (9.1) [lower limit 9.1] | -74.4 (6.3) [lower limit 6.3]

15. Secondary Outcome: Absolute Change in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Week 24 (ITT Estimand)
Description: Absolute change in non-HDL-C from baseline at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
mg/dL | -0.4 (17.4) [lower limit 17.4] | -148.0 (12.3) [lower limit 12.3]

16. Secondary Outcome: Absolute Change in Total Cholesterol (TC) From Baseline to Week 24 (ITT Estimand)
Description: Absolute change in TC from baseline at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
mg/dL | -0.4 (17.2) [lower limit 17.2] | -161.6 (12.2) [lower limit 12.2]

17. Secondary Outcome: Percent Change in Apolipoprotein CIII (Apo CIII) From Baseline to Week 24 (ITT Estimand)
Description: Percent change in Apo CIII from baseline at Week 24 in the DBTP was reported; value obtained regardless of adherence to study treatment and subsequent therapies (ITT estimand). ITT population included all randomized participants who received at least one dose or part of a dose of double-blind study drug. Participants in the ITT population were analyzed according to the treatment group allocated by randomization (i.e., as randomized participant group).
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo IV Q4W | Evinacumab 15 mg/kg IV Q4W
Number analyzed (Participants) | 22 | 43
Percent Change | 5.8 (5.5) [lower limit 5.5] | -84.1 (3.9) [lower limit 3.9]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up until end of study (Week 68) regardless of seriousness or relationship to investigational product (IP).
Description: For purpose of safety analysis, arm assignments for participants in Safety Set were based on actual treatment received, such that 1 participant assigned to Placebo arm who inadvertently received evinacumab 15mg/kg was included in Evinacumab 15mg/kg arm
Arm/Group | Placebo IV Q4W (DBTP) | Evinacumab 15 mg/kg (DBTP) | Placebo IV Q4W (OLTP) | Evinacumab 15 mg/kg (OLTP)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/44 | 0/20 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/44 | 0/20 | 7/44
Other Adverse Events (participants affected / at risk) | 13/21 | 20/44 | 12/20 | 19/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV Q4W (DBTP) (N=21) | Evinacumab 15 mg/kg (DBTP) (N=44) | Placebo IV Q4W (OLTP) (N=20) | Evinacumab 15 mg/kg (OLTP) (N=44)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo IV Q4W (DBTP) (N=21) | Evinacumab 15 mg/kg (DBTP) (N=44) | Placebo IV Q4W (OLTP) (N=20) | Evinacumab 15 mg/kg (OLTP) (N=44)
Nasopharyngitis (Infections and infestations) | 5 (6) | 7 (7) | 1 (2) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (8) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 4 (7) | 1 (2) | 5 (5)
Influenza like illness (General disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menstrual discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03399786/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT03399786/SAP_001.pdf